CLINICAL TRIAL: NCT01324479
Title: A Phase I Open-label Dose Escalation Study With Expansion to Assess the Safety and Tolerability of INC280 in Patients With c-MET Dependent Advanced Solid Tumors
Brief Title: Study of INC280 in Patients With c-MET Dependent Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC280X2102; 2010-024101-12 (EudraCT Number)
Record Dates: First submitted 2011-03-25; First posted 2011-03-29 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2019-04

CONDITIONS: Solid Tumors
Keywords: Non-small cell lung cancer,; hepatocellular,; gastric,; renal cell,; c-MET,; refractory,; glioblastoma,; breast,; nasopharyngeal,; confirmed evidence of c-MET dysregulation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Glioblastoma | interventions — capmatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INC280 (Experimental)
  Interventions: Drug: INC280

INTERVENTIONS:
Drug: INC280

SUMMARY:
This study will assess the safety and efficacy of INC280 in patients with solid tumors that are refractory to current treatment or for which there is not a current standard of care and whose tumors have dysregulation of the c-MET pathway.

ELIGIBILITY:
Inclusion Criteria:

* Must have evidence of c-MET dysregulation from either local data or the results of molecular pre-screening evaluations.
* Confirmed diagnosis of a solid tumor.
* Measureable lesion.
* Refractory to currently available treatment or no therapies available.
* 18 years or older.
* ECOG performance status of 0, 1, or 2.
* Obtained written informed consent.

Additional inclusion criteria for NSCLC patients EGFRwt with high c-MET expression:

* Written documentation of EGFRwt NSCLC.
* Written documentation of c-MET positivity.
* Patients should not have received more than three prior lines of antineoplastic therapy for NSCLC.
* Presence of at least one measurable lesion as determined by modified RECIST version 1.1

Exclusion Criteria:

HCC with liver dysfunction greater than Child-Pugh A. Previous treatment with a c-MET inhibitor or HGF-targeting therapy. Symptomatic CNS metastases that are neurologically unstable or requiring increasing doses of steroids to control their CNS disease.

Any CNS deficits. For patients with GBM, CNS symptoms grade 2 or greater. Subjects with significant or uncontrolled cardiovascular disease (eg, uncontrolled hypertension, peripheral vascular disease, congestive heart failure, cardiac arrhythmia, or acute coronary syndrome) within 6 months of starting study treatment or heart attack within 12 months of starting study treatment.

Receiving anti-epileptic drugs that are known to be strong inducers of CYP3A4. Prior or current anti-angiogenic therapy for patients with GBM. Radiation therapy within ≤ 4 weeks (< 12 for GBM) prior to the first dose of study drug or limited field radiotherapy within ≤ 2 weeks (< 12 weeks GBM) prior to the start of study treatment. Any persistent side effect of prior radiotherapy must be resolved to ≤ Grade 1 prior to the first dose of study drug.

Additional exclusion criteria for NSCLC patients EGFRwt with high c-MET expression:

* Patients who have received more than three prior lines of antineoplastic therapies
* Any unresolved toxicity (CTCAE grade > 1) from previous anti-cancer therapy or radiotherapy, except alopecia
* Patients have received anti-cancer therapies within the following time frames prior to the first dose of study treatment:

  * Conventional cytotoxic chemotherapy: ≤4 weeks (≤6 weeks for nitrosoureas and mitomycin-C)
  * Biologic therapy (e.g., antibodies): ≤4 weeks
  * Non-cytotoxic small molecule therapeutics: ≤5 half-lives or ≤2 weeks (whichever is longer)
  * Other investigational agents: ≤4 weeks
  * Radiation therapy (palliative setting is allowed.): ≤4 weeks
  * Major surgery: ≤2 weeks

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2012-02-29 (Actual); Primary Completion 2017-07-04 (Actual); Study Completion 2017-07-04 (Actual)

PRIMARY OUTCOMES:
Incidence rate of dose-limiting toxicities and adverse events | 2 years

SECONDARY OUTCOMES:
Objective response by local investigator assessment | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (45):
- United States (5):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - University of Chicago SC, Chicago, Illinois
  - Karmanos Cancer Institute Wayne St Karmanos, Detroit, Michigan
  - Sarah Cannon Research Institute Dept of Onc, Nashville, Tennessee
  - University of Texas/MD Anderson Cancer Center Dept of Onc, Houston, Texas
- Australia (2):
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Woolloongabba, Queensland
- Canada (2):
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
- France (3):
  - Novartis Investigative Site, La Tronche
  - Novartis Investigative Site, Lille Cédex
  - Novartis Investigative Site, Strasbourg
- Germany (6):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Oldenburg
- Hong Kong (2):
  - Novartis Investigative Site, Shatin, New Territories, Hong Kong
  - Novartis Investigative Site, Hong Kong
- Israel (4):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (4):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Meldola, FC
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Reggio Emilia, RE
- Netherlands (3):
  - Novartis Investigative Site, Utrecht, The Netherlands
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Rotterdam
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Singapore, Singapore
- South Korea (4):
  - Novartis Investigative Site, Seoul, Gyeonggi-do
  - Novartis Investigative Site, Gyeonggi-do, Korea
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seocho Gu
- Spain (5):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Zaragoza
- Taiwan (2):
  - Novartis Investigative Site, Tainan, Taiwan ROC
  - Novartis Investigative Site, Taipei, Taiwan ROC
- Novartis Investigative Site, Songkhla, Hat Yai, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schuler M, Berardi R, Lim WT, de Jonge M, Bauer TM, Azaro A, Gottfried M, Han JY, Lee DH, Wollner M, Hong DS, Vogel A, Delmonte A, Akimov M, Ghebremariam S, Cui X, Nwana N, Giovannini M, Kim TM. Molecular correlates of response to capmatinib in advanced non-small-cell lung cancer: clinical and biomarker results from a phase I trial. Ann Oncol. 2020 Jun;31(6):789-797. doi: 10.1016/j.annonc.2020.03.293. Epub 2020 Mar 30. PMID 32240796
- [Derived] Bang YJ, Su WC, Schuler M, Nam DH, Lim WT, Bauer TM, Azaro A, Poon RTP, Hong D, Lin CC, Akimov M, Ghebremariam S, Zhao S, Giovannini M, Ma B. Phase 1 study of capmatinib in MET-positive solid tumor patients: Dose escalation and expansion of selected cohorts. Cancer Sci. 2020 Feb;111(2):536-547. doi: 10.1111/cas.14254. Epub 2019 Dec 30. PMID 31778267
- See also: Results for INC280X2102 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17178